CLINICAL TRIAL: NCT01998854
Title: Observational Prospective Study on Patients With Symptomatic Uterine Fibroids Treated With VizAblate® Intrauterine-ultrasound Guided RF Ablation
Status: Terminated | Type: Observational
Why Stopped: Investigational device changes
Sponsor: Gynesonics (Industry)
Responsible Party: Sponsor
Other Study IDs: CL03537
Record Dates: First submitted 2013-11-25; First posted 2013-12-02 (Estimated); Last update posted 2015-03-11 (Estimated); Status verified 2015-03

CONDITIONS: Menorrhagia; Leiomyoma; Uterine Fibroids; Uterine Fibroma; Uterine Neoplasms
Keywords: Menorrhagia; Leiomyoma; Uterine Fibroids
MeSH Terms: conditions — Menorrhagia; Leiomyoma; Uterine Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- VizAblate treatment: VizAblate System with subject serving as her own control
  Interventions: Device: VizAblate System

INTERVENTIONS:
Device: VizAblate System — The VizAblate System is indicated for use in transcervical intrauterine-guided radio frequency ablation of uterine fibroids

SUMMARY:
Study is intended to evaluate the one-year safety and clinical status of patients treated for symptomatic uterine fibroids with the VizAblate Intrauterine-ultrasound guided radio frequency (RF) ablation system. Particular attention will be directed to recording safety outcomes including incidence of uterine cavity synechiae. In addition, information on quality of life will be collected.

Overall study duration (first patient enrolled through last patient exit) will be comprised of approximately 12 months of patient enrollment up to 1 month for scheduling of treatment, and 12 months of follow-up, for a total duration of up to 25 months. Study duration for an individual patient, once enrolled, will be approximately 1 month for baseline observations and treatment scheduling, and 12 months for follow up after treatment for a total duration of approximately 13 months.

DETAILED DESCRIPTION:
In this single-arm study, subjects who receive transcervical intrauterine-ultrasound guided RF ablation of symptomatic uterine fibroids with the VizAblate® System will be assessed with 3D pelvic sonography with contrast, hysteroscopy, and quality of life questionnaires.

Overall study duration (first patient enrolled through last patient exit) will be comprised of approximately 12 months of patient enrollment up to 1 month for scheduling of treatment, and 12 months of follow-up, for a total duration of up to 25 months. Study duration for an individual patient, once enrolled, will be approximately 1 month for baseline observations and treatment scheduling, and 12 months for follow up after treatment for a total duration of approximately 13 months.

ELIGIBILITY:
Inclusion Criteria:

* 28 years of age or older
* Indication for transcervical treatment of uterine fibroids associated with menorrhagia
* Willingness to participate in the study, to attend all follow-up visits and undergo all study assessments, and to sign the informed consent form
* Presence of submucosal and/or intramural fibroids

Exclusion Criteria:

* Pregnancy
* ≥40 years of age with desire for current or future fertility, unless the estimated risk/benefit ratio has been determined to be more favorable to future pregnancy than standard therapy
* Non-sterilized patients < 40 years of age, unless the estimated risk/benefit ratio has been determined to be more favorable to future pregnancy than standard therapy
* Active pelvic infection, known or suspected gynecologic malignancy or premalignant condition
* Presence of tubal implant for sterilization
* Previous pelvic irradiation
* Endometrial cavity length, including endocervical canal, < 4.5 cm
* Any abnormality of the vagina or uterine cavity that, in the judgment of the investigator obstructs access of the VizAblate handpiece to the endometrial cavity
* Presence of cardiac pacemaker or other active implant
* Post-menopausal

Min Age: 28 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients of specified clinical sites with complaint of symptomatic uterine fibroids.
Sampling Method: Non-Probability Sample
Enrollment: 4 (Actual)
Dates: Start 2013-02; Primary Completion 2014-06 (Actual); Study Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
Mean percentage change in treated fibroid perfused volume | 12 months

SECONDARY OUTCOMES:
Fibroid total volume reduction | 12 months
Incidence of Intrauterine adhesiogenesis | 7 weeks
  The cavity will be as classified per the European Society for Hysteroscopy (ESH)
Procedure Safety | Day of procedure
  Frequency and type of adverse events occurring on the day of the procedure
Long-term safety | 12 months
  Frequency and type of adverse events occurring post treatment through 12 months
Percentage reduction in the Symptom Severity Score sub scale of the Uterine Fibroid Symptom - Quality of Life questionnaire | 12 months
Percentage increase in the Health Related Quality-of-Life (HRQL) sub scale of the Uterine Fibroid Symptom-Quality of Life questionnaire | 12 months
Rate of surgical reintervention for menorrhagia | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: David Toub, MD, Study Director — Gynesonics
Locations (2):
- France (2):
  - Le Centre Hospitalier Regional et Universitaire de Tours - Hôpital Bretonneau, Tours, Cedex
  - Assistance Publique Hôpitaux de Paris - Hôpital Bicêtre, Paris